CLINICAL TRIAL: NCT02813941
Title: Two Alternatives Versus Usual GRADE-SoF Tables to Improve Understanding in the Presentation of Systematic Review Results: A Three-arm, Randomized, Controlled, Noninferiority Trial
Brief Title: Comparison of Three Summary of Finding Tables to Improve Understanding in the Presentation of Systematic Review Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Grading of Recommendations Assessment, Development and Evaluation working group (Unknown); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MIF1-II; NCT02732028 (obsolete NCT alias)
Record Dates: First submitted 2016-06-20; First posted 2016-06-27 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Research Report
Keywords: Randomized controlled trial; Systematic review; Summary of finding tables; GRADE; AHRQ

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alternative GRADE SoF table (Experimental): Two SoF tables (alternative GRADE SoF table and EPC SoF table) will be used in this randomized controlled non-inferiority trial as an intervention. The alternative GRADE SoF table format will be developed from a user-testing survey.
  Interventions: Other: Current GRADE SoF table
- EPC SoF table (Experimental): For the EPC SoF table, the investigators will use one of their format which was recently published.
  Interventions: Other: Alternative GRADE SoF table
- Current GRADE SoF table (Active Comparator): The current GRADE SoF table will be the common comparator for the other two SoF tables
  Interventions: Other: EPC SoF table

INTERVENTIONS:
Other: Current GRADE SoF table — The current GRADE SoF table will be the common comparator for the other two SoF tables
  Other Names: Table A
  Arms: Alternative GRADE SoF table
Other: Alternative GRADE SoF table — The alternative GRADE SoF table format will be developed from a user-testing survey.
  Other Names: Table B
  Arms: EPC SoF table
Other: EPC SoF table — For the EPC SoF table, the investigators will use one of their format which was recently published
  Other Names: Table C
  Arms: Current GRADE SoF table

SUMMARY:
Background: Summary of Findings (SoF) tables have been developed to present results of systematic reviews in a concise and explicit format. Adopted by many review groups including the Cochrane Collaboration, the Agency for Healthcare Research and Quality (AHRQ), and the GRADE Working Group; SoF tables provide succinct, transparent, and easily interpretable judgments about the certainty of evidence and magnitude of effects. Currently, there are three different SoF formats in use. This study aims to compare SoF table formats in terms of understanding, accessibility, satisfaction, and preference with systematic review users.

Methods: The primary objective of this three-arm randomized controlled non-inferiority trial is to investigate whether an alternative GRADE-SoF table, or EPC-SoF table, is noninferior to the current GRADE-SoF table in the understanding of information presented to systematic review users. Researchers, clinical practice guideline developers, policy-makers, end-users, or knowledge transfer will be recruited. Data will be collected electronically at baseline and after randomization. Noninferiority would be declared if the difference in the proportion of participants who understand the information displayed in the alternative SoF table is 10% or less.

Discussion: This study aims to assess the understanding, accessibility, satisfaction, and preference between three SoF tables for displaying summary evidence from health-related outcomes. The results of this study will provide important knowledge to understand what information should be included in SoF tables in systematic reviews.

DETAILED DESCRIPTION:
Objective: Summary of Findings (SoF) tables present results of systematic reviews in a concise and explicit format. Adopted by many review groups including the Cochrane Collaboration, and the Agency for Healthcare Research and Quality (AHRQ). Optimal understanding of SoF table may be influenced by the type of information being conveyed and objectives or preferences of the end user. This study aims to compare three SoF table formats in terms of understanding, accessibility, satisfaction, and preference with systematic review users.

Methods: The primary objective of this three-arm randomized controlled non-inferiority trial is to investigate whether an alternative GRADE-SoF table or EPC-SoF table is noninferior to the current GRADE-SoF table in the understanding of the information presented to systematic review users, particularly for descriptive findings. Researchers, clinical practice guideline developers, policy-makers, or knowledge transfer professionals will be recruited. Data will be collected electronically at baseline and after randomization. Noninferiority would be declared if the difference in the proportion of participants who understand the information displayed in the alternative SoF table is 10% or less.

Ethics and Dissemination: The Hamilton Integrated Research Ethics Board (HiREB) reviewed this protocol. The findings from this study will be disseminated through a publication in a peer-reviewed journal.

Strengths and limitations of this study

* This is a randomized controlled trial that uses a GRADE Summary of Finding (SoF) table evaluated in another randomized controlled trial with a positive accomplishment of understanding the information displayed on it.
* This is the first time that GRADE SoF tables will be evaluated, in terms of understanding descriptive findings with a select part of a SoF table adapted by an EPC center to convey information on multiple comparisons efficiently.
* This will test understanding of presentation of findings from only a single comparison and will not test understanding of a complex body of evidence.

ELIGIBILITY:
Inclusion criteria:

Participants will be eligible if they consider themselves as systematic review users. For the purpose of this trial, systematic review users will be defined as researchers, clinical practice guideline developers, policy-makers, or knowledge transfer professionals. Participants who declare dedicating more than 70% of their time during last year to conducting research (for example, methodologists, epidemiologists, statisticians) will be classified as researchers. Participants who declare having participated in at least one systematic review or clinical practice guideline during the last two years will be classified as clinical practice guideline developers. Knowledge transfer professionals, who declare working in a dynamic and iterative process that includes synthesis, dissemination, exchange and ethically sound application of knowledge to improve the health care system, during last two years, will be classified as knowledge transfer professionals. Finally, participants who declare being responsible for or involved in formulating policies in the last year, especially in politics, will be classified as policy-makers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Understanding of information (questionnaire) | 30 minutes
  Investigators will frame multiple-choice questions about key concepts in the table with five response alternatives for each question and only one correct answer. Then, investigators will compare the proportion of correct answers between groups per question

SECONDARY OUTCOMES:
Accessibility of information (questionnaire) | 30 minutes
  This outcome considers four items: 1) how easy it is to find critical information in the table; 2) how easy it is to understand the information; 3) whether the information is presented in a way that is helpful for decision-making; and 4) the overall accessibility of information.
Satisfaction (questionnaire) | 30 minutes
  It will be measured using a 7-point Likert scale with 3 anchors: 1= strongly dissatisfied, 4= neither satisfied nor dissatisfied, 7= strongly satisfied, and it will be treated as a continuous outcome. Investigators will compare the means per group.
Preference (questionnaire) | 30 minutes
  Participants will answer the question: 'Between Table A (the current GRADE SoF table), Table B (the alternative GRADE SoF table) or Table C (EPC SoF table), which table do you prefer?' It will be measured using a rank of three: 1st choice, 2nd choice, and 3rd choice, and it will be treated as an ordinal outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Holger J Schunemann, MD, MSc, PhD, Principal Investigator — McMaster University, Department of Clinical Epidemiology & Biostatistics
Locations (1):
- Department of Health Research Methods, Evidence and Impact, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There will be no individual patient data shared from this study.

REFERENCES:
- [Result] Berkman ND, Lohr KN, Ansari MT, Balk EM, Kane R, McDonagh M, Morton SC, Viswanathan M, Bass EB, Butler M, Gartlehner G, Hartling L, McPheeters M, Morgan LC, Reston J, Sista P, Whitlock E, Chang S. Grading the strength of a body of evidence when assessing health care interventions: an EPC update. J Clin Epidemiol. 2015 Nov;68(11):1312-24. doi: 10.1016/j.jclinepi.2014.11.023. Epub 2014 Dec 20. PMID 25721570
- [Result] Feltner C, Jones CD, Cene CW, Zheng ZJ, Sueta CA, Coker-Schwimmer EJL, Arvanitis M, Lohr KN, Middleton JC, Jonas DE. Transitional Care Interventions To Prevent Readmissions for People With Heart Failure [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 May. Report No.: 14-EHC021-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK209241/ PMID 24967474
- [Result] Carrasco-Labra A, Brignardello-Petersen R, Santesso N, Neumann I, Mustafa RA, Mbuagbaw L, Etxeandia Ikobaltzeta I, De Stio C, McCullagh LJ, Alonso-Coello P, Meerpohl JJ, Vandvik PO, Brozek JL, Akl EA, Bossuyt P, Churchill R, Glenton C, Rosenbaum S, Tugwell P, Welch V, Garner P, Guyatt G, Schunemann HJ. Improving GRADE evidence tables part 1: a randomized trial shows improved understanding of content in summary of findings tables with a new format. J Clin Epidemiol. 2016 Jun;74:7-18. doi: 10.1016/j.jclinepi.2015.12.007. Epub 2016 Jan 11. PMID 26791430
- [Derived] Yepes-Nunez JJ, Morgan RL, Mbuagbaw L, Carrasco-Labra A, Chang S, Hempel S, Shekelle P, Helfand M, Baldeh T, Schunemann HJ. Two alternatives versus the standard Grading of Recommendations Assessment, Development and Evaluation (GRADE) summary of findings (SoF) tables to improve understanding in the presentation of systematic review results: a three-arm, randomised, controlled, non-inferiority trial. BMJ Open. 2018 Jan 23;8(1):e015623. doi: 10.1136/bmjopen-2016-015623. PMID 29362242
- See also: Online survey — https://www.surveymonkey.com